CLINICAL TRIAL: NCT04604990
Title: National Systemic Lupus Erythematosus Prospective Cohort, Saudi Arabia
Status: Recruiting | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ibrahim Almaghlouth, Principle Investigator, King Saud University
Other Study IDs: E-19-3955/8
Record Dates: First submitted 2020-10-12; First posted 2020-10-27 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: SLE (Systemic Lupus)
Keywords: SLE; Lupus erythematosus; Outcomes; Phenotypes; Observational
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each patient will have two comprehensive visit during which 4 heparin blood tubes will be collected from the patient for biobanking storage (exception will be for pregnant patients who will have biological sample collection at the beginning of each trimester along with postpartum sample (six weeks from delivery).
  Once the blood is withdrawn, it will be sorted into:
  plasma separation, (immune cell sorting using flow cytometry to into major cell line including T-cells, B cells, mononuclear cells and granulocytes/versus storage as PBMC - the decision will be guided by available fund), RNA and DNA then stored at appropriate temperature using patient unique research identification number.
  For DNA processing; blood will be collected using standardized phlebotomy technique directly into PAXgene Blood DNA tubes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SLE disease in Saudi Arabia is yet not well defined especially in a population with high consanguinity and high inbreeding coefficient . Up until now, there has been no prospective cohort study for SLE patients in Saudi Arabia. As a result, current published literature is focused on retrospective chart reviews which are subjected to many forms of bias. so the investigator proposed this prospective registry which will follow open cohort study design aiming to provide better understanding of disease presentation, course and outcomes especially if complemented by detailed immunological, molecular, genetic and microbiome data.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients defined as age greater than 18 years old.
2. Patients should fulfil one of the following classification criteria for SLE (ACR, SLICC or ACR/EULAR criteria).
3. No restriction on time of diagnosis.

Exclusion Criteria:

* Patients who don't fulfil classification criteria mentioned above.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from KSU-SLE specialized clinic. The clinic receive general referral from general rheumatology clinics in KSU and general referral from other clinics inside or outside KSU. The estimated number is 1000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2050-11-01 (Estimated); Study Completion 2050-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease Accrual damage among SLE patients in Saudi Arabia | over 10 years
  SLEDAI-2K, Systemic Lupus Erythematosus Disease Activity Index 2000 (0-150) higher score representing higher disease activity
Disease Accrual damage among SLE patients in Saudi Arabia | over 10 years
  SLICC/ACR DI, Systemic Lupus International Collaboration Clinics/ American College of Rheumatology
Disease Accrual damage among SLE patients in Saudi Arabia | over 10 years
  Mortality

SECONDARY OUTCOMES:
Patient reported outcome | over 5 years
  PROMIS ( Patient Reported Outcome Measurement Information Scale) there are several data collection tool for calculating score (will use REDCap auto score). Each question usually has 5 response option ranging in value from one to five. For example, the adult 8-item, the lowest possible score is 8, the highest possible score is 40
Patient reported outcome | over 5 years
  Medication adherence by using Modified Medication Adherence Response Scale (Modified MARS), an overall score of 4 and above is considered adherent.
Fetal and maternal outcomes in patients with SLE | over 5 years
  Intrauterine fetal death, Abortion, Still birth, Eclampsia and pre-eclampsia, disease Activity

CONTACTS AND LOCATIONS:
Locations (1):
- king Saud University medical city, Riyadh, Central Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF
Time Frame: upon recruitment, informed consent form will be shared and before enrolment.

REFERENCES:
- [Derived] Almaghlouth IA, Hassen LM, Alahmari HS, Bedaiwi A, Albarrak R, Daghestani M, Alqurtas E, Alkhalaf A, Bedaiwi M, Omair M, Almogairen S, Alarfaj H, Alarfaj A. National systemic lupus erythematosus prospective cohort in Saudi Arabia: A study protocol. Medicine (Baltimore). 2021 Jul 30;100(30):e26704. doi: 10.1097/MD.0000000000026704. Erratum In: Medicine (Baltimore). 2021 Aug 27;100(34):e27039. doi: 10.1097/MD.0000000000027039. PMID 34397699

DOCUMENTS (1):
  • Study Protocol (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04604990/Prot_000.pdf